CLINICAL TRIAL: NCT03696862
Title: Assessment of Collagen Plug Versus Free Gingival Graft for Alveolar Socket Sealing With Simultaneous Implant Placement in Maxillary Esthetic Zone
Brief Title: Assessment of Collagen Plug for Alveolar Socket Sealing With Simultaneous Implant Placement in Maxillary Esthetic Zone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, sara elsandouby, principal investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CairoUimplant master porgram
Record Dates: First submitted 2018-09-16; First posted 2018-10-05 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Badly Decayed Upper Anterior Teeth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- collagen plug (Experimental): collagen plug used to seal the socket after atraumatic extraction of the badly deacayed teeth with immediate implant placement and bone graft
  Interventions: Procedure: free gingival graft

INTERVENTIONS:
Procedure: free gingival graft — Use of free gingival graft to seal the socket after flapless atraumatic tooth extraction is performed, implant placement and filling the socket with bone graft.

SUMMARY:
Following tooth extraction alveolar ridge will undergo dimensional changes and soft tissue may collapse. These changes may complicate the subsequent restorative procedure especially in the esthetic zone.

It was observed that socket-healing process may be divided into three sequential, and frequently over-lapping phases: inflammatory, proliferative and modeling/remodeling.

Implants placed in fresh extraction sockets alone wasn't found to prevent the resorption of the alveolar bone.

DETAILED DESCRIPTION:
Alveolar socket preservation using primary flap closure technique utilizing free gingival graft in conjunction with bone substitutes didn't produce the desired effect on ridge preservation compared with bone substitutes alone. A clinical trial showed that achieving primary closure didn't present additional beneficial effect on preserving ridge width, however, the mucosa was significantly thicker and more coronally positioned.

Also soft tissue graft has its limitations on covering graft material and socket preservation due to the higher morbidity given that the soft tissue graft has to be harvested from a donor site of the patient.

Another options for socket seal are coronal advancement of buccal flap or rotating grafts from tissue adjacent to cover the defect but they have limitations such as altering the mucogingival line and creating a shallow vestibule.

Lekovic et al. investigated the use of a non-resorbable polytetrafluroethylene membrane but it was found also to have its limitations as 30% of the membranes became exposed and as a result loss of bone height and width occurred.

Also studies have found that using bone substitutes together with collagen membrane with primary closure of the socket has shown clear effects on preserving alveolar ridge height as well as ridge width, however, its limitation are flap dehiscence and subsequent membrane exposure and the increased cost.

ELIGIBILITY:
Inclusion Criteria:

* Patients with maxillary teeth in the esthetic zone (incisors/premolars) requiring extractions.
* Both sexes.
* No intraoral soft and hard tissue pathology.
* No systemic condition that contraindicate implant placement.

Exclusion Criteria:

* Uncontrolled periapical infections
* Heavy smokers more than 20 cigarettes per day.
* Patients with systemic disease that may affect normal healing.
* Psychiatric problems
* Disorders to implant are related to history of radiation therapy to the head and neck neoplasia, or bone augmentation to implant site
* Immunodeficiency pathology, bruxism, stress situation (socially or professionally), emotional instability, and unrealistic aesthetic demands.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-10-20 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
changes in soft tissue | 3 month
  soft tissue changes will be measured in millimeters clinically and on a cast before and after the procedure
changes in bone | 6 month
  bone loss and gain will be measured in millimeters using cone beam computed tomography before and after the procedure